CLINICAL TRIAL: NCT06642402
Title: Monitoring and Detecting Lupus Nephritis Through Urinary Extracellular Vesicles in Urine
Brief Title: Monitoring Lupus Nephritis Through Urinary Extracellular Vesicles
Status: Recruiting | Type: Observational
Sponsor: Kolding Sygehus (Other)
Collaborators: University of Southern Denmark (Other); Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SLELNuEV
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus Nephritis
Keywords: Systemic Lupus Erythoematosus nephritis; Lupus nephritis; complement activation; kidney biopsy
MeSH Terms: conditions — Lupus Nephritis | interventions — Autoimmunity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Detailed demographic and clinical data including age, sex, ethnicity, medicine, duration of SLE activity, SLE damage and laboratory results will be collected from each patient.
  Blood samples will be collected and tested for immun markers of lupus nephritis.
  Urine samples willl be collected to detect kidney function and to isolate urinary extracellular vesicles.
  Kidney biopsies will be histological analyzed at department of Pathology by experienced nephro-pathologists according to existing clinical guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Systemic lupus erythomatosus with lupus nephritis: SLE patients with kidney involvement
  Interventions: Diagnostic Test: Kidney biopsy; Diagnostic Test: Urinary extracellular vesicle testing; Diagnostic Test: Autoimmunity in plasma
- Systemic lupus erythomatosus without lupus nephritis: SLE patients, fulfilling the 2019 EULAR/ACR classification criteria with no sign of kidney disease
  Interventions: Diagnostic Test: Urinary extracellular vesicle testing; Diagnostic Test: Autoimmunity in plasma
- Healthy controls: Healthy controls
  Interventions: Diagnostic Test: Urinary extracellular vesicle testing
- Biopsy controls: A biopsy control group with no predictive complement activation referred to biopsy
  Interventions: Diagnostic Test: Kidney biopsy; Diagnostic Test: Urinary extracellular vesicle testing

INTERVENTIONS:
Diagnostic Test: Kidney biopsy — Patient refered to kidney biopsy independent of the presented study
  Other Names: No expected complement activation
  Groups: Biopsy controls; Systemic lupus erythomatosus with lupus nephritis
Diagnostic Test: Urinary extracellular vesicle testing — Urinary extracellular vesicles will be isolated and tested for complement activation and other markers of kidney disease
Diagnostic Test: Autoimmunity in plasma — Expected autoimmunity in plasma isolated from blood samples
  Groups: Systemic lupus erythomatosus with lupus nephritis; Systemic lupus erythomatosus without lupus nephritis

SUMMARY:
Lupus nephritis (LN) is a severe manifestation of systemic lupus erythematosus (SLE) that can lead to irreversible kidney damage if not detected and managed promptly. LN is classified and treated based on its histopathological features obtained by invasive kidney biopsy. Recent research has suggested urinary extracellular vesicles (uEVs) as potential non-invasive biomarkers. The primary objective of this prospective study is to investigate the utility of uEVs in LN.

DETAILED DESCRIPTION:
Introduction: Lupus nephritis (LN) is a severe manifestation of systemic lupus erythematosus (SLE) that can lead to irreversible kidney damage if not detected and managed promptly. LN is classified based on its histopathological features. The classification helps in determining the severity and appropriate treatment strategies for the condition and to rule out other conditions that may mimic the clinical picture of LN. The classification system most commonly used is the International Society of Nephrology/Renal Pathology Society (ISN/RPS) classification, which divides lupus nephritis into six classes: I) Minimal Change, II) Mesangial Proliferative LN, III) Focal Proliferative LN, IV) Diffus proliferative LN, V) Membranous LN, VI) Advanced Sclerosing LN. The classification requires invasive kidney biopsies, which are hardly accessible and associated with potential complications and patient discomfort. Furthermore the kidney biopsy only represent a small part of the kidney. Recent research has suggested urinary extracellular vesicles (uEVs) as potential non-invasive biomarkers for kidney diseases, including LN. uEVS are small nano-sized extracellular vesicles of endosomal origin, which are secreted into the urine through fusion of multivesicular bodies with the plasma membrane. Thus, they could represent a promising liquid biopsy that reflects the pattern and/or severity of renal injury.

Hypothesis: The primary objective of this prospective study is to investigate the utility of urinary exosomes as non-invasive biomarkers for monitoring the activity and progression of lupus nephritis.

Methods: SLE patients, fulfilling the 2019 EULAR/ACR classification criteria, referred to kidney biopsy, will be recruited from Department of Rheumatology and Department of Nephrology at Odense University Hospital. Detailed demographic and clinical data including age, sex, ethnicity, medicine, duration of SLE activity, SLE damage and laboratory results will be collected from each patient. Activity of SLE at the time of biopsy will be evaluated using SLE disease activity index 2000 (SLEDAI-2K). SLE damage will be evaluated in accordance with the SLICC damage index. Spot-urine samples will be collected, added protease-inhibitors and frozen at -80 degree. UEVs will be isolated using polyethylene glycol (PEG) precipitation, the concentration of uEV will be determined and protein accessed using western blotting and/or PCR. Glomerular specific uEVs will be isolated and previous developed tests will be applied to detect the membrane attack complex (MAC)/C5b-9 complex. uEVs from plasma/serum will be isolated to test for correlation with uEVs. Kidney biopsies will be histological analyzed at Department of Pathology by experienced nephropathologists according to existing clinical guidelines. Differences in uEV cargo between SLE patients with and without lupus nephritis will be analyzed using appropriate statistical tests. Correlations between uEV biomarkers, histological differences on the kidney biopsy and disease activity will be evaluated using Pearson's correlation analysis.

Perspective: This prospective study aims to establish urinary extracellular vesicles as potential non-invasive biomarkers for monitoring lupus nephritis in SLE patients. The findings from this research may lead to the development of more efficient and patient-friendly approaches for LN management, enabling timely interventions and improved renal outcomes in SLE patients.

ELIGIBILITY:
SLE patients with kidney involvement

Inclusion criteria:

* > 18 years old
* Fulfilling the 2019 EULAR/ACR classification criteria
* Positive autoantibodies, medical history and obejctive examination compatible with SLE
* Referred to kidney biopsy

Exclusion criteria:

* Lack of ability or willingness to provide informed consent
* Significant comorbidity, which is considered to potentially impact the outcome

SLE patients with no sign of kidney disease

Inclusion criteria:

* > 18 years old
* Fulfilling the 2019 EULAR/ACR classification criteria
* Positive autoantibodies, medical history and obejctive examination compatible with SLE
* Normal plasma creatinine
* Urine albumine/creatinine < 100 mg/g

Exclusion criteria:

* Lack of ability or willingness to provide informed consent
* Significant comorbidity, which is considered to potentially impact the outcome

Healthy controls:

Inclusion criteria:

* > 18 years old
* No known kidney disease

Exclusion criteria:

* Lack of ability or willingness to provide informed consent
* Urine albumin-creatinine ratio > 100 mg/g or proteinuria > 100 mg/day
* Postive autoantibodies
* Significant comorbidity, which is considered to potentially impact the outcome

Biopsy control:

Inclusion criteria:

* > 18 years old
* Negative autoantibiodies and immunoglobulines
* Referred to kidney biopsy

Exclusion criteria:

* Lack of ability or willingness to provide informed consent
* Significant comorbidity, which is considered to potentially impact the outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients known with SLE with and without kidney involvement, a biopsy control and a group of healthy controls.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between kidney biopsy and urinay extracellular vesicles | Urinary extracellular vesicles will be isolated from urine collected at the day of kidney biopsy/baseline. Analysis will be performed when all samples are collected. Estimated after 5 years.
  The primary outcome is to investigate the correlation between histological findings from kidney biopsy and urinary extracelluar vesicles, with the aim of assessing whether there is concordance between the two methods in relation to disease severity and classification.
Complement activation in urinary extracellular vesicles | Measured on urinary extracellular vesicles obtained at the day of biopsy/baseline. Analysis will be performed when all samples are collected, estimated after 5 years.
  Urinary extracellular vesicles will be isolated. Complement activation will be detected using an in-house ELISA assay

SECONDARY OUTCOMES:
Correlation between urinary extracellular vesicles and extracellular vesicles from plasma | Blood- og and urine samples will be collected at the day of kidney biopsy/baseline. Analysis will be performed when all samples are collecting, estimated after 5 years.
  A seconday outcome is to invesigate the correlation between urinary extracellular vesicles and extracellular vesicles from plasma, to see if the same results could be obtained in plasma samples

CONTACTS AND LOCATIONS:
Overall Officials: Anne F Christensen, Chief of Medicine, MD, phd, Study Chair — Sygehus Lillebaelt, Kolding Hospitl
Locations (4):
- Denmark (4):
  - Kolding Hospital, Kolding
  - Department of Nephrology, Odense
  - Department of Rheumatology, Odense
  - Univesity of Southern Denmark, Odense

IPD SHARING:
Plan to Share IPD: Undecided